CLINICAL TRIAL: NCT06961331
Title: Real-world Clinical Outcomes of Tucatinib, Trastuzumab, and Capecitabine Following Trastuzumab Deruxtecan for the Treatment of HER2-postive Metastatic Breast Cancer
Brief Title: Real World-clinical Outcomes of Tucatinib, Trastuzumab, and Capecitabine Following Trastuzumab Deruxtecan (T-DXd) for the Treatment of HER2-positive Metastatic Breast Cancer.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4251025
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic HER2+ Advanced Breast Cancer
Keywords: her2+; mBC; metastatic breast cancer; tukysa; tucatinib; breast neoplasm; Human epidermal growth factor receptor 2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- 3L+4L tucatinib triplet patients: Non-interventional, retrospective cohort analysis of participants receiving the tucatinib triplet in the 3L or 4L setting immediately following T-DXd.
  Interventions: Drug: Tucatinib; Drug: Trastuzumab; Drug: Capecitabine

INTERVENTIONS:
Drug: Tucatinib — As provided in real world practice.
Drug: Trastuzumab — As provided in real world practice.
Drug: Capecitabine — As provided in real world practice.

SUMMARY:
A retrospective study of de-identified (to preserve patient privacy) patient information from the Flatiron Health Database to describe 3L and 4L real-world (rw) outcomes (e.g. time to next treatment, time to discontinuation, and overal survival) of the tucatinib-trastuzumab-capecitabine triplet therapy immediately following T-DXd therapy in patients diagnosed with HER2+ metastatic breast cancer (mBC) in the United States.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. mBC diagnosis between January 1, 2017 and 6 months prior to database cutoff
2. Evidence of human epidermal growth factor receptor 2 (HER2) receptor positivity prior to or up to 90 days following the mBC diagnosis date
3. At least 18 years old on the mBC diagnosis date
4. Treated with systemic anticancer treatment in the metastatic setting, i.e., post mBC diagnosis.
5. Treated with T-DXd in the 1L or 2L or 3L setting, followed immediately by the tucatinib triplet, and at least 1 additional prior HER2-targeted regimen

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Patients with evidence of other cancers six months prior to the mBC diagnosis date will be identified with the following International Classification of Diseases, 9th Revision, Clinical Modification (ICD-9-CM) and International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) codes in all databases: 140.xx - 195.xx, 200.xx - 208.xx, C00.xx - C76.xx, C81.xx - C96.xx. (exclude - ICD-9: 174.X, 175.X; ICD-10: C50.XX)
2. Patients treated with tucatinib prior to T-DXd
3. Patients participating in clinical trials
4. Patients receiving concomitant endocrine therapy on index line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include participants in the US Flatiron Dataset diagnosed with HER2+ mBC treated with the tucatinib triplet in the post-T-DXd setting.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Time to Next Treatment | 1 Year
  Time to next treatment defined as the time in months from the initiation of therapy to the initiation of subsequent LOT or death.
Time to Discontinuation | 1 Year
  Time to treatment discontinuation defined as the time in months from initiation of therapy to discontinuation for any reason or death.
Overall survival (OS) | 1 Year
  OS will be defined as the time in months from initiation of therapy to death from any cause.
real-world Progression free survival (rwPFS) | 1 Year
  rwPFS will be defined as time in months from initiation of therapy to progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4251025